CLINICAL TRIAL: NCT01411228
Title: A Multicenter Extension Study of Taliglucerase Alfa in Pediatric Subjects With Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PB-06-006
Expanded Access: NCT00962260 (No longer available)
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; pediatrics
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 60 Units/kg (Experimental)
  Interventions: Drug: Taliglucerase alfa
- 30 Units/kg (Experimental)
  Interventions: Drug: Taliglucerase alfa

INTERVENTIONS:
Drug: Taliglucerase alfa — Taliglucerase alfa for infusion every two weeks for 24 months
  Other Names: prGCD, plant cell expressed glucocerebrosidase

SUMMARY:
A protocol to extend the assessment of the safety and efficacy of taliglucerase alfa in pediatric subjects (2 to <18 years old) with symptoms and clinical manifestations of Gaucher disease who completed treatment in Protocols PB-06-002 (switchover study from imiglucerase) or PB-06-005 (naïve treatment with taliglucerase alfa).

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of Protocol PB-06-002 or PB-06-005
* The subject, parent(s) or legal guardian(s) signs an informed consent and/or assent

Exclusion Criteria:

* Currently taking another investigational drug for any condition.
* Presence of neurological signs and symptoms characteristic of Gaucher disease with complex neuronopathic features other than longstanding oculomotor gaze palsy.
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the subject's compliance with the requirements of the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Shaare Zedek Medical Center, Jerusalem, Israel
- Instituto Privado de Hematologia E Investigacion Clinica (I.P.H.I.C), Barrio Asunción, Paraguay
- Morningside Medi-Clinic, Morningside, South Africa

REFERENCES:
- [Derived] Zimran A, Gonzalez-Rodriguez DE, Abrahamov A, Cooper PA, Varughese S, Giraldo P, Petakov M, Tan ES, Chertkoff R. Long-term safety and efficacy of taliglucerase alfa in pediatric Gaucher disease patients who were treatment-naive or previously treated with imiglucerase. Blood Cells Mol Dis. 2018 Feb;68:163-172. doi: 10.1016/j.bcmd.2016.10.005. Epub 2016 Oct 20. PMID 27839981
- [Derived] Abbas R, Park G, Damle B, Chertkoff R, Alon S. Pharmacokinetics of Novel Plant Cell-Expressed Taliglucerase Alfa in Adult and Pediatric Patients with Gaucher Disease. PLoS One. 2015 Jun 8;10(6):e0128986. doi: 10.1371/journal.pone.0128986. eCollection 2015. PMID 26053270

RESULTS

PARTICIPANT FLOW:
Groups:
- Switchover: Taliglucerase alfa: Taliglucerase alfa for infusion every two weeks for 24 months
Period: Overall Study
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Started | 5 | 5 | 5
Completed | 4 | 5 | 4
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Adjusted: Taliglucerase alfa: Dose increased from 30 Units/kg to 45 or 60 Units/kg
- Total: Total of all reporting groups
Arm/Group | 60 Units/kg | 30 Units/kg | Dose Adjusted | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (3.1) | 8.6 (3.8) | 13.0 (4.1) | 9.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 4 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 2 | 1 | 0 | 3
  Israel | 2 | 1 | 0 | 3
  Spain | 0 | 0 | 2 | 2
  Serbia | 0 | 0 | 2 | 2
  Paraguay | 1 | 3 | 0 | 4
  Singapore | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin
Description: Median and interquartile range. Baseline is the value obtained from the parent study: PB-06-005 for 30 and 60 Units/kg arms and PB-06-002 from Switchover arm.
Time Frame: Baseline, months 9, 12 and 24
Population: Two Switchover Patients completed 18 months treatment due to early closure of the study site and continued in a compassionate use program
Measure: Median (Inter-Quartile Range); unit: g/dL
Groups:
- Switchover: Taliglucerase alfa: Maintained dose from PB-06-002 study
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Number analyzed (Participants) | 5 | 5 | 5
g/dL
  Baseline | 10.6 [9.1 to 12.3] | 11.2 [9.1 to 12.3] | 13.5 [12.9 to 14.2]
  Month 9 | 11.9 [10.5 to 13.8] | 12.5 [10.1 to 13.7] | 13.9 [12.5 to 15.2]
  Month 12 | 12.2 [11.2 to 13.7] | 12.8 [11.2 to 14.2] | 13.7 [12.0 to 15.1]
  Month 24 | 12.8 [11.0 to 14.2] | 13.1 [11.5 to 14.5] | 14.2 [12.1 to 16.0]

2. Secondary Outcome: Chitotriosidase
Description: Chitotriosidase. Baseline is the value obtained from the parent study: PB-06-005 for 30 and 60 Units/kg arms and PB-06-002 from Switchover arm.
Time Frame: Baseline, months 9, 12 and 24
Population: Chitotriosidase was not analyzed for the subjects in the Switchover group
Measure: Mean (Standard Deviation); unit: nmol/mL*h
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Number analyzed (Participants) | 5 | 4 | 0
nmol/mL*h
  Baseline | 34968 (20928) | 30783 (17771) |
  Month 9 | 17416 (16821) | 13983 (10562) |
  Month 12 | 14677 (14418) | 13823 (11525) |
  Month 24 | 7449.5 (6966.5) | 10079 (9452.4) |

3. Secondary Outcome: Spleen Volume
Description: Spleen volume measured by MRI (or ultrasound). Baseline is the value obtained from the parent study: PB-06-005 for 30 and 60 Units/kg arms and PB-06-002 from Switchover arm.
Time Frame: Baseline, months 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Milliliters
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Number analyzed (Participants) | 5 | 5 | 5
Milliliters
  Baseline | 1023.1 (336.9) | 1244.7 (317.6) | 313.0 (69.8)
  12 Months | 524.0 (125.7) | 759.0 (194.4) | 274.1 (39.3)
  24 Months | 395.8 (76.8) | 719.0 (161.2) | 249.5 (69.8)
  33-36 Months | 306.1 (55.1) | 673.2 (128.7) | 185.4 (12.6)

4. Secondary Outcome: Platelet Count
Description: Platelet count. Baseline is the value obtained from the parent study: PB-06-005 for 30 and 60 Units/kg arms and PB-06-002 from Switchover arm.
Time Frame: Baseline, months 9, 12, 24 and 33-36
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Platelets/mm^3
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Number analyzed (Participants) | 5 | 5 | 5
Platelets/mm^3
  Baseline | 99600 (19185) | 182000 (27009) | 164587 (17321)
  Month 9 | 172600 (38667) | 221400 (30626) | 177400 (16795)
  Month 12 | 172200 (39932) | 233800 (32759) | 189000 (7733.0)
  Month 24 | 192800 (26673) | 207600 (18291) | 234800 (14867)
  Month 33-36 | 243750 (18585) | 220200 (29231) | 210000 (10000)

5. Secondary Outcome: Liver Volume
Description: Liver volume by MRI or Ultrasound. Baseline is the value obtained from the parent study: PB-06-005 for 30 and 60 Units/kg arms and PB-06-002 from Switchover arm.
Time Frame: Baseline, months 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Milliliters
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Number analyzed (Participants) | 5 | 5 | 5
Milliliters
  Baseline | 991.7 (134.7) | 1236.5 (210.6) | 1345.6 (193.1)
  Month 12 | 849.1 (121.6) | 1140.6 (180.9) | 1460.7 (227.8)
  Month 24 | 865.5 (82.4) | 1254.4 (114.9) | 1480.7 (253.3)
  Month 33-36 | 890.6 (118.2) | 1244.8 (89.1) | 1274.2 (189.7)

ADVERSE EVENTS:
Arm/Group | 60 Units/kg | 30 Units/kg | Switchover
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 Units/kg (N=5) | 30 Units/kg (N=5) | Switchover (N=5)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — (Grade 2 Dengue Fever), which required hospitalization, resolved in 5 weeks and was assessed as not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 Units/kg (N=5) | 30 Units/kg (N=5) | Switchover (N=5)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
DENGUE FEVER (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No